CLINICAL TRIAL: NCT04198402
Title: Microbiotic Analysis in Digestive Endocrine Tumors
Acronym: MicroTEND
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190427
Record Dates: First submitted 2019-12-04; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-11

CONDITIONS: Digestive Neuroendocrine Tumor; Fecal Microbiota; Bacterial Signature

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fecal sample blood sample
  blood sample is part of routine medical care and fecal sample is a non invasive collection of elements from human body, allowing the study to be categorised as a non-interventional research (approved by ethics commitee)
  Please see:
  "Arrêté du 12 avril 2018 fixant la liste des recherches mentionnées au 3° de l'article L. 1121-1 du code de la santé publique" , justifying observational study type
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with digestive neuroendocrine tumor: naive patient with digestive neuroendocrine tumor (pancreas or small intestine), initiating Lanreotide treatment
  Interventions: Biological: Biological sampling
- Patient without tumor: Historical control group (retrospective data) Patients, with normal endoscopic and body imaging results, having had fecal ARN16s sequencing who were assigned as control subjects for microbiota analyses.

INTERVENTIONS:
Biological: Biological sampling — Blood sample (5mL) for metabolomic dosage and Fecal sample for ARN16s sequencing
  Groups: Patient with digestive neuroendocrine tumor

SUMMARY:
Incidence of digestive neuroendocrine tumors are increasing. Analysis of individual microbiota is a way to explore new neoplastic mechanisms, tumor identification and therapeutic orientations. This prospective pilot study aims to describe fecal bacterial phylogeny of patients with digestive neuroendocrine tumor.

Bacterial genomic signature will be recorded at initiation of Lanreotide treatment in naive patient with digestive neuroendocrine tumor (pancreas or small intestine), metastatic or locally advanced, as well as after one year follow up.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* naive patient with digestive neuroendocrine tumor (pancreas (cytology or histology per endoscopy or on surgical specimen) or small intestine), secreting or not, initiating a extended release Lanreotide treatment
* registered with a social security scheme

Exclusion Criteria:

* medical contraindication to somatostatine analogs use
* history of extended release somatostatine analogs treatment
* antibiotic use or colonoscopic purge in the last 3 weeks preceding fecal sample
* pregnant or breastfeeding women
* person requiring tutorship, guardianship, or person legally protected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Naive patient with digestive neuroendocrine tumor (pancreas (cytology or histology per endoscopy or on surgical specimen) or small intestine), secreting or not, going to receive Lanreotide treatment as the first line therapy for their disease.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
bacterial genomic signature | Baseline visit
  bacterial genomic signature by fecal ARN16S analysis at enrollment

IPD SHARING:
Plan to Share IPD: No
Data are own by Assistance Publique - Hopitaux de Paris, please contact sponsor for further information